CLINICAL TRIAL: NCT05746767
Title: SUPERA: Supporting Peer Interactions to Expand Access to Digital Cognitive Behavioral Therapy for Spanish-speaking Safety-Net Patients in Primary Care
Brief Title: Supporting Peer Interactions to Expand Access to Digital Cognitive Behavioral Therapy for Spanish-speaking Patients
Acronym: SUPERA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Berkeley (Other); University of California, San Francisco (Other); University of California, Riverside (Other); University of New Mexico (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Stephen Matthew Schueller, Professor of Psychological Science, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1856; R01MH126664 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Depression, Anxiety
Keywords: Digital Health Intervention; Mobile Health; Digital Cognitive-Behavioral Therapy; Peer Supporter
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Comparing peer-supported delivery vs. unsupported delivery of dCBT
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants randomly assigned to this condition will be provided all features of the SilverCloud platform as well as be assigned a peer-supporter who will provide regular support.
  Interventions: Behavioral: Supported dCBT
- Control (Active Comparator): Participants randomly assigned to this condition will be provided all features of the SilverCloud platform with the exception of the peer supporter.
  Interventions: Behavioral: Unsupported dCBT

INTERVENTIONS:
Behavioral: Supported dCBT — In the supported dCBT condition, each patient will receive complete access to the SilverCloud platform. In addition, patients will be assigned a supporter who will provide regular support based on an established coaching support protocol. Supporters will conduct a brief engagement call (30-40 minutes) to provide an overview of SilverCloud, identify goals, and set expectations, introduce themselves, and orient the participant to the role of the peer supporter. Supporters will then provide weekly check-ins through phone calls or messaging. Participants will be able to communicate with the supporters through the platform through messaging or sharing activities for additional discussion. The major goal of the support is to promote use of the platform.
  Arms: Treatment
Behavioral: Unsupported dCBT — Unsupported dCBT provides all features of the SilverCloud platform with the exception of support features (structured interactions with supporter and share features). Patients will be provided complete access to SilverCloud and instructed to use it for 8-weeks. Patients will receive weekly automated messages to encourage engagement.
  Arms: Control

SUMMARY:
Investigators will evaluate the implementation of an evidence-based, Spanish-language, digital, cognitive-behavioral therapy intervention (SilverCloud) in primary care settings for Latino patients with depression and/or anxiety. 426 participants will be enrolled in a two-armed trial comparing self-guided vs. supported dCBT (SilverCloud). At the provider level, investigators will compare the efficacy of provider referrals with the use of a clinic patient registry to identify candidates who could benefit from a digital mental health intervention.

DETAILED DESCRIPTION:
The investigators will evaluate the implementation of an evidence-based, Spanish language, digital cognitive-behavioral therapy (dCBT) intervention (SilverCloud) in safety-net primary care clinics for Limited English Proficiency (LEP) Latinx patients with depression and/or anxiety. An effectiveness-implementation hybrid trial (Type 2) design with patient-level randomization. The implementation comparison will evaluate a non-randomized comparison between outreach (using the clinic patient registry) with inreach (traditional provider referral). The effectiveness comparison will include randomization at the patient-level to two modes of delivery of the dCBT platform - supported and unsupported will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. PHQ-9 ≥ 10 or GAD-7 ≥ 8
2. Has access to the Internet via smartphone and/or broadband at home, and basic level of technological literacy or willingness to undergo a brief technology use training
3. ≥18 years of age
4. Preference for receiving medical care in Spanish
5. Not in concurrent psychotherapy
6. If currently taking an antidepressant medication, patient must have been on a stable dose for at least 6 weeks, and have no plans to change the dose. We will permit patients on antidepressants to enter the study, as this will increase generalizability. Antidepressant status will be monitored at each assessment to control for those effects, if necessary.

Exclusion Criteria:

1. Currently receiving psychotherapy, as this treatment will be offered as a frontline treatment for depression and anxiety, however, patients are allowed to be referred to treatment while participating in this study and initiation of treatment will be monitored and considered in analyses
2. Visual, hearing, voice, or motor impairment or illiteracy that would prevent completion of study procedures
3. Diagnosis of a psychotic disorder, bipolar disorder, dissociative disorder, or substance use disorder
4. Severe suicidality (as assessed by expressing suicidal ideation, plan, and intent). Although procedures with back-up plans are in place for patients who develop suicidality (see Human Subjects Section), patients assessed with severe suicidality will be referred to more-intensive treatment resources.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depression at 8 Weeks | Change from Baseline to Week 8
  The primary outcome of symptoms of depression will be measured with the self-report Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report measure of depression. Scores on this measure range from 0 (Not At All) to 3 (Nearly Every Day).
Change in Anxiety at 8 Weeks | Change from Baseline to Week 8
  The primary outcome of symptoms of depression will be measured with the self-report General Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item self-report measure of anxiety. Scores on this measure range from 0 (Not At All) to 3 (Nearly Every Day).

SECONDARY OUTCOMES:
Change in Functioning at 8 Weeks | Change from Baseline to Week 8
  Functioning will be assessed with the World Health Organization Disability Assessment Schedule (WHODAS) a 36-item self-report measure that assesses disability across six domains, including understanding and communicating, getting around, self-care, getting along with people, life activities (i.e., household, work, and/or school activities), and participation in society. Scores on this measure range from 1 (none) to 5 (extreme).
Platform Usage | Total platform usage from baseline to Week 8
  Platform usage will be defined as time spent on the platform. Platform usage will vary from 0 minutes to the highest number of minutes any participants spends on the platform.

OTHER OUTCOMES:
Change in Frequency of Applying CBT-Based Skills at 8 Weeks | Change from Baseline to Week 8
  Frequency of Actions and Thoughts Scale (FATS). A 12-item measure that will be used to assess how frequently the participants apply CBT-based skills. Higher score means that the respondent has higher frequency of applying the CBT-based skills they learned.
Change in Knowledge of CBT at 8 Weeks | Change from Baseline to Week 8
  Knowledge Gain in CBT. A 16-item survey that will be used to assess changes in knowledge about CBT therapy. Higher score means that the respondent has higher knowledge of CBT skills.
Change in Psychological Well-Being | Change from Baseline to Week 8
  Psychological Well-Being will be assessed with the Brief Inventory of Thriving (BIT) a 10-item self-report measure. Scores on this measure range from 5 (low level of thriving) to 50 (high level of thriving).
Change in Stress at 8 Weeks | Change from Baseline to Week 8
  Stress will be assessed with the Perceived Stress Scale (PSS-4) a 4-item self-report measure that assesses feelings and thoughts that people are experiencing related to their experience of stress. Scores on this measure range from 0 (no perceived stress) to 16 (high perceived stress).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Schueller, PhD, Principal Investigator — University of California, Irvine; Adrian Aguilera, PhD, Principal Investigator — University of California, Berkeley
Locations (11):
- United States (11):
  - Payson Christian Clinic, Payson, Arizona
  - Family and Community Medicine Mobile Health Clinic, Tucson, Arizona
  - University of California, Berkeley, California
  - University of California, Irvine, California
  - Zuckerberg San Francisco General, San Francisco, California
  - Castro-Mission Health Center, San Francisco, California
  - Silver Avenue Family Health Center, San Francisco, California
  - UNMH North Valley Clinic, Albuquerque, New Mexico
  - Truman Health Clinic, Albuquerque, New Mexico
  - UNM Southeast Heights Clinic, Albuquerque, New Mexico
  - Sandoval Regional Medical Center, Rio Rancho, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be deposited in a NIH data repository the NIMH Data Archive
Time Frame: Descriptive data will be submitted every six months. Analyzed datasets on study outcomes will be deposited in the repository as soon as possible but no later than within one year of the completion of the project. No end date on data availability.
Access Criteria: Anyone who wishes to access the data and adheres to the NIMH Data Archive policies.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Gonzalez JM, Alegria M, Prihoda TJ, Copeland LA, Zeber JE. How the relationship of attitudes toward mental health treatment and service use differs by age, gender, ethnicity/race and education. Soc Psychiatry Psychiatr Epidemiol. 2011 Jan;46(1):45-57. doi: 10.1007/s00127-009-0168-4. Epub 2009 Nov 17. PMID 19921079
- [Background] Falgas I, Ramos Z, Herrera L, Qureshi A, Chavez L, Bonal C, McPeck S, Wang Y, Cook B, Alegria M. Barriers to and Correlates of Retention in Behavioral Health Treatment Among Latinos in 2 Different Host Countries: The United States and Spain. J Public Health Manag Pract. 2017 Jan/Feb;23(1):e20-e27. doi: 10.1097/PHH.0000000000000391. PMID 26910867
- [Background] Kim G, Aguado Loi CX, Chiriboga DA, Jang Y, Parmelee P, Allen RS. Limited English proficiency as a barrier to mental health service use: a study of Latino and Asian immigrants with psychiatric disorders. J Psychiatr Res. 2011 Jan;45(1):104-10. doi: 10.1016/j.jpsychires.2010.04.031. Epub 2010 May 26. PMID 20537658
- [Background] Sentell T, Shumway M, Snowden L. Access to mental health treatment by English language proficiency and race/ethnicity. J Gen Intern Med. 2007 Nov;22 Suppl 2(Suppl 2):289-93. doi: 10.1007/s11606-007-0345-7. Epub 2007 Oct 24. PMID 17957413
- [Background] Bauer AM, Chen CN, Alegria M. English language proficiency and mental health service use among Latino and Asian Americans with mental disorders. Med Care. 2010 Dec;48(12):1097-104. doi: 10.1097/MLR.0b013e3181f80749. PMID 21063226
- [Background] Kazdin AE, Blase SL. Rebooting Psychotherapy Research and Practice to Reduce the Burden of Mental Illness. Perspect Psychol Sci. 2011 Jan;6(1):21-37. doi: 10.1177/1745691610393527. Epub 2011 Feb 3. PMID 26162113
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] National Collaborating Centre for Mental Health (UK). Depression: The Treatment and Management of Depression in Adults (Updated Edition). Leicester (UK): British Psychological Society; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK63748/ PMID 22132433
- [Background] Gilbody S, Littlewood E, Hewitt C, Brierley G, Tharmanathan P, Araya R, Barkham M, Bower P, Cooper C, Gask L, Kessler D, Lester H, Lovell K, Parry G, Richards DA, Andersen P, Brabyn S, Knowles S, Shepherd C, Tallon D, White D; REEACT Team. Computerised cognitive behaviour therapy (cCBT) as treatment for depression in primary care (REEACT trial): large scale pragmatic randomised controlled trial. BMJ. 2015 Nov 11;351:h5627. doi: 10.1136/bmj.h5627. PMID 26559241
- [Background] Graham AK, Lattie EG, Powell BJ, Lyon AR, Smith JD, Schueller SM, Stadnick NA, Brown CH, Mohr DC. Implementation strategies for digital mental health interventions in health care settings. Am Psychol. 2020 Nov;75(8):1080-1092. doi: 10.1037/amp0000686. PMID 33252946
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Vilsaint CL, NeMoyer A, Fillbrunn M, Sadikova E, Kessler RC, Sampson NA, Alvarez K, Green JG, McLaughlin KA, Chen R, Williams DR, Jackson JS, Alegria M. Racial/ethnic differences in 12-month prevalence and persistence of mood, anxiety, and substance use disorders: Variation by nativity and socioeconomic status. Compr Psychiatry. 2019 Feb;89:52-60. doi: 10.1016/j.comppsych.2018.12.008. Epub 2018 Dec 19. PMID 30594752
- [Background] Escovar EL, Craske M, Roy-Byrne P, Stein MB, Sullivan G, Sherbourne CD, Bystritsky A, Chavira DA. Cultural influences on mental health symptoms in a primary care sample of Latinx patients. J Anxiety Disord. 2018 Apr;55:39-47. doi: 10.1016/j.janxdis.2018.03.005. Epub 2018 Mar 12. PMID 29576380
- [Background] Wells K, Klap R, Koike A, Sherbourne C. Ethnic disparities in unmet need for alcoholism, drug abuse, and mental health care. Am J Psychiatry. 2001 Dec;158(12):2027-32. doi: 10.1176/appi.ajp.158.12.2027. PMID 11729020
- [Background] Brody DS, Khaliq AA, Thompson TL 2nd. Patients' perspectives on the management of emotional distress in primary care settings. J Gen Intern Med. 1997 Jul;12(7):403-6. doi: 10.1046/j.1525-1497.1997.00070.x. PMID 9229277
- [Background] Dwight-Johnson M, Sherbourne CD, Liao D, Wells KB. Treatment preferences among depressed primary care patients. J Gen Intern Med. 2000 Aug;15(8):527-34. doi: 10.1046/j.1525-1497.2000.08035.x. PMID 10940143
- [Background] Bedi N, Chilvers C, Churchill R, Dewey M, Duggan C, Fielding K, Gretton V, Miller P, Harrison G, Lee A, Williams I. Assessing effectiveness of treatment of depression in primary care. Partially randomised preference trial. Br J Psychiatry. 2000 Oct;177:312-8. doi: 10.1192/bjp.177.4.312. PMID 11116771
- [Background] Priest RG, Vize C, Roberts A, Roberts M, Tylee A. Lay people's attitudes to treatment of depression: results of opinion poll for Defeat Depression Campaign just before its launch. BMJ. 1996 Oct 5;313(7061):858-9. doi: 10.1136/bmj.313.7061.858. PMID 8870574
- [Background] Churchill R, Khaira M, Gretton V, Chilvers C, Dewey M, Duggan C, Lee A; Nottingham Counselling and Antidepressants in Primary Care (CAPC) Study Group. Treating depression in general practice: factors affecting patients' treatment preferences. Br J Gen Pract. 2000 Nov;50(460):905-6. PMID 11141877
- [Background] Givens JL, Houston TK, Van Voorhees BW, Ford DE, Cooper LA. Ethnicity and preferences for depression treatment. Gen Hosp Psychiatry. 2007 May-Jun;29(3):182-91. doi: 10.1016/j.genhosppsych.2006.11.002. PMID 17484934
- [Background] Interian A, Ang A, Gara MA, Rodriguez MA, Vega WA. The long-term trajectory of depression among Latinos in primary care and its relationship to depression care disparities. Gen Hosp Psychiatry. 2011 Mar-Apr;33(2):94-101. doi: 10.1016/j.genhosppsych.2010.12.001. Epub 2011 Jan 19. PMID 21596201
- [Background] Chavira DA, Golinelli D, Sherbourne C, Stein MB, Sullivan G, Bystritsky A, Rose RD, Lang AJ, Campbell-Sills L, Welch S, Bumgardner K, Glenn D, Barrios V, Roy-Byrne P, Craske M. Treatment engagement and response to CBT among Latinos with anxiety disorders in primary care. J Consult Clin Psychol. 2014 Jun;82(3):392-403. doi: 10.1037/a0036365. Epub 2014 Mar 24. PMID 24660674
- [Background] Forde F, Frame M, Hanlon P, MacLean G, Nolan D, Shajahan P, Troy E. Optimum number of sessions for depression and anxiety. Nurs Times. 2005 Oct 25-31;101(43):36-40. PMID 16276843
- [Background] Hansen NB, Lambert MJ. An evaluation of the dose-response relationship in naturalistic treatment settings using survival analysis. Ment Health Serv Res. 2003 Mar;5(1):1-12. doi: 10.1023/a:1021751307358. PMID 12602642
- [Background] Nieuwsma JA, Trivedi RB, McDuffie J, Kronish I, Benjamin D, Williams JW. Brief psychotherapy for depression: a systematic review and meta-analysis. Int J Psychiatry Med. 2012;43(2):129-51. doi: 10.2190/PM.43.2.c. PMID 22849036
- [Background] Frank RG, Huskamp HA, Pincus HA. Aligning incentives in the treatment of depression in primary care with evidence-based practice. Psychiatr Serv. 2003 May;54(5):682-7. doi: 10.1176/appi.ps.54.5.682. PMID 12719498
- [Background] Dwight-Johnson M, Lagomasino IT, Hay J, Zhang L, Tang L, Green JM, Duan N. Effectiveness of collaborative care in addressing depression treatment preferences among low-income Latinos. Psychiatr Serv. 2010 Nov;61(11):1112-8. doi: 10.1176/ps.2010.61.11.1112. PMID 21041350
- [Background] Olfson M, Blanco C, Marcus SC. Treatment of Adult Depression in the United States. JAMA Intern Med. 2016 Oct 1;176(10):1482-1491. doi: 10.1001/jamainternmed.2016.5057. Erratum In: JAMA Intern Med. 2016 Oct 1;176(10):1579. doi: 10.1001/jamainternmed.2016.6486. PMID 27571438
- [Background] Horevitz E, Organista KC, Arean PA. Depression Treatment Uptake in Integrated Primary Care: How a "Warm Handoff" and Other Factors Affect Decision Making by Latinos. Psychiatr Serv. 2015 Aug 1;66(8):824-30. doi: 10.1176/appi.ps.201400085. Epub 2015 Apr 15. PMID 25873022
- [Background] Yabroff KR, O'Malley A, Mangan P, Mandelblatt J. Inreach and outreach interventions to improve mammography use. J Am Med Womens Assoc (1972). 2001 Fall;56(4):166-73, 188. PMID 11759785
- [Background] Fuzzell LN, Perkins RB, Christy SM, Lake PW, Vadaparampil ST. Cervical cancer screening in the United States: Challenges and potential solutions for underscreened groups. Prev Med. 2021 Mar;144:106400. doi: 10.1016/j.ypmed.2020.106400. Epub 2021 Jan 1. PMID 33388330
- [Background] Guendelman S, Witt S. Improving access to prenatal care for latina immigrants in california: outreach and inreach strategies. Int Q Community Health Educ. 1991 Jan 1;12(2):89-106. doi: 10.2190/HV3W-JD07-1Y7L-N3N5. PMID 20840961
- [Background] Becker SJ. Direct-to-Consumer Marketing: A Complementary Approach to Traditional Dissemination and implementation Efforts for Mental Health and Substance Abuse Interventions. Clin Psychol (New York). 2015 Mar 1;22(1):85-100. doi: 10.1111/cpsp.12086. PMID 25937710
- [Background] Karyotaki E, Efthimiou O, Miguel C, Bermpohl FMG, Furukawa TA, Cuijpers P; Individual Patient Data Meta-Analyses for Depression (IPDMA-DE) Collaboration; Riper H, Patel V, Mira A, Gemmil AW, Yeung AS, Lange A, Williams AD, Mackinnon A, Geraedts A, van Straten A, Meyer B, Bjorkelund C, Knaevelsrud C, Beevers CG, Botella C, Strunk DR, Mohr DC, Ebert DD, Kessler D, Richards D, Littlewood E, Forsell E, Feng F, Wang F, Andersson G, Hadjistavropoulos H, Christensen H, Ezawa ID, Choi I, Rosso IM, Klein JP, Shumake J, Garcia-Campayo J, Milgrom J, Smith J, Montero-Marin J, Newby JM, Breton-Lopez J, Schneider J, Vernmark K, Bucker L, Sheeber LB, Warmerdam L, Farrer L, Heinrich M, Huibers MJH, Kivi M, Kraepelien M, Forand NR, Pugh N, Lindefors N, Lintvedt O, Zagorscak P, Carlbring P, Phillips R, Johansson R, Kessler RC, Brabyn S, Perini S, Rauch SL, Gilbody S, Moritz S, Berger T, Pop V, Kaldo V, Spek V, Forsell Y. Internet-Based Cognitive Behavioral Therapy for Depression: A Systematic Review and Individual Patient Data Network Meta-analysis. JAMA Psychiatry. 2021 Apr 1;78(4):361-371. doi: 10.1001/jamapsychiatry.2020.4364. PMID 33471111
- [Background] Graham AK, Greene CJ, Kwasny MJ, Kaiser SM, Lieponis P, Powell T, Mohr DC. Coached Mobile App Platform for the Treatment of Depression and Anxiety Among Primary Care Patients: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Sep 1;77(9):906-914. doi: 10.1001/jamapsychiatry.2020.1011. PMID 32432695
- [Background] Titov N, Dear BF, Staples LG, Bennett-Levy J, Klein B, Rapee RM, Andersson G, Purtell C, Bezuidenhout G, Nielssen OB. The first 30 months of the MindSpot Clinic: Evaluation of a national e-mental health service against project objectives. Aust N Z J Psychiatry. 2017 Dec;51(12):1227-1239. doi: 10.1177/0004867416671598. Epub 2016 Oct 12. PMID 27733709
- [Background] Titov N, Dear B, Nielssen O, Staples L, Hadjistavropoulos H, Nugent M, Adlam K, Nordgreen T, Bruvik KH, Hovland A, Repal A, Mathiasen K, Kraepelien M, Blom K, Svanborg C, Lindefors N, Kaldo V. ICBT in routine care: A descriptive analysis of successful clinics in five countries. Internet Interv. 2018 Jul 26;13:108-115. doi: 10.1016/j.invent.2018.07.006. eCollection 2018 Sep. PMID 30206525
- [Background] Duffy D, Enrique A, Connell S, Connolly C, Richards D. Internet-Delivered Cognitive Behavior Therapy as a Prequel to Face-To-Face Therapy for Depression and Anxiety: A Naturalistic Observation. Front Psychiatry. 2020 Jan 9;10:902. doi: 10.3389/fpsyt.2019.00902. eCollection 2019. PMID 31998149
- [Background] Moberg C, Niles A, Beermann D. Guided Self-Help Works: Randomized Waitlist Controlled Trial of Pacifica, a Mobile App Integrating Cognitive Behavioral Therapy and Mindfulness for Stress, Anxiety, and Depression. J Med Internet Res. 2019 Jun 8;21(6):e12556. doi: 10.2196/12556. PMID 31199319
- [Background] Dryman MT, McTeague LM, Olino TM, Heimberg RG. Evaluation of an open-access CBT-based Internet program for social anxiety: Patterns of use, retention, and outcomes. J Consult Clin Psychol. 2017 Oct;85(10):988-999. doi: 10.1037/ccp0000232. Epub 2017 Jun 26. PMID 28650193
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885
- [Background] Richards D, Enrique A, Eilert N, Franklin M, Palacios J, Duffy D, Earley C, Chapman J, Jell G, Sollesse S, Timulak L. Erratum: Author Correction: A pragmatic randomized waitlist-controlled effectiveness and cost-effectiveness trial of digital interventions for depression and anxiety. NPJ Digit Med. 2020 Jun 30;3:91. doi: 10.1038/s41746-020-0298-3. eCollection 2020. PMID 32637656
- [Background] Salamanca-Sanabria A, Richards D, Timulak L. Adapting an internet-delivered intervention for depression for a Colombian college student population: An illustration of an integrative empirical approach. Internet Interv. 2019 Jan 14;15:76-86. doi: 10.1016/j.invent.2018.11.005. eCollection 2019 Mar. PMID 30740313
- [Background] Salamanca-Sanabria A, Richards D, Timulak L, Connell S, Mojica Perilla M, Parra-Villa Y, Castro-Camacho L. A Culturally Adapted Cognitive Behavioral Internet-Delivered Intervention for Depressive Symptoms: Randomized Controlled Trial. JMIR Ment Health. 2020 Jan 31;7(1):e13392. doi: 10.2196/13392. PMID 32003749
- [Background] Titov N, Andrews G, Davies M, McIntyre K, Robinson E, Solley K. Internet treatment for depression: a randomized controlled trial comparing clinician vs. technician assistance. PLoS One. 2010 Jun 8;5(6):e10939. doi: 10.1371/journal.pone.0010939. PMID 20544030
- [Background] Aguilera A, Garza MJ, Munoz RF. Group cognitive-behavioral therapy for depression in Spanish: culture-sensitive manualized treatment in practice. J Clin Psychol. 2010 Aug;66(8):857-67. doi: 10.1002/jclp.20706. PMID 20549680
- [Background] Barnett ML, Gonzalez A, Miranda J, Chavira DA, Lau AS. Mobilizing Community Health Workers to Address Mental Health Disparities for Underserved Populations: A Systematic Review. Adm Policy Ment Health. 2018 Mar;45(2):195-211. doi: 10.1007/s10488-017-0815-0. PMID 28730278
- [Background] Hoeft TJ, Fortney JC, Patel V, Unutzer J. Task-Sharing Approaches to Improve Mental Health Care in Rural and Other Low-Resource Settings: A Systematic Review. J Rural Health. 2018 Dec;34(1):48-62. doi: 10.1111/jrh.12229. Epub 2017 Jan 13. PMID 28084667
- [Background] Waitzkin H, Getrich C, Heying S, Rodriguez L, Parmar A, Willging C, Yager J, Santos R. Promotoras as mental health practitioners in primary care: a multi-method study of an intervention to address contextual sources of depression. J Community Health. 2011 Apr;36(2):316-31. doi: 10.1007/s10900-010-9313-y. PMID 20882400
- [Background] Schueller SM, Aguilera A, Mohr DC. Ecological momentary interventions for depression and anxiety. Depress Anxiety. 2017 Jun;34(6):540-545. doi: 10.1002/da.22649. Epub 2017 May 11. PMID 28494123
- [Background] Mohr DC, Lyon AR, Lattie EG, Reddy M, Schueller SM. Accelerating Digital Mental Health Research From Early Design and Creation to Successful Implementation and Sustainment. J Med Internet Res. 2017 May 10;19(5):e153. doi: 10.2196/jmir.7725. PMID 28490417
- [Background] Aarons GA, Sklar M, Mustanski B, Benbow N, Brown CH. "Scaling-out" evidence-based interventions to new populations or new health care delivery systems. Implement Sci. 2017 Sep 6;12(1):111. doi: 10.1186/s13012-017-0640-6. PMID 28877746
- [Background] Aguilera A, Schueller SM, Leykin Y. Daily mood ratings via text message as a proxy for clinic based depression assessment. J Affect Disord. 2015 Apr 1;175:471-4. doi: 10.1016/j.jad.2015.01.033. Epub 2015 Jan 29. PMID 25679202
- [Background] Bruehlman-Senecal E, Aguilera A, Schueller SM. Mobile Phone-Based Mood Ratings Prospectively Predict Psychotherapy Attendance. Behav Ther. 2017 Sep;48(5):614-623. doi: 10.1016/j.beth.2017.01.002. Epub 2017 Jan 9. PMID 28711112
- [Background] Aguilera A, Munoz RF. Text Messaging as an Adjunct to CBT in Low-Income Populations: A Usability and Feasibility Pilot Study. Prof Psychol Res Pr. 2011 Dec 1;42(6):472-478. doi: 10.1037/a0025499. PMID 25525292
- [Background] Aguilera A, Berridge C. Qualitative feedback from a text messaging intervention for depression: benefits, drawbacks, and cultural differences. JMIR Mhealth Uhealth. 2014 Nov 5;2(4):e46. doi: 10.2196/mhealth.3660. PMID 25373390
- [Background] Aguilera A, Bruehlman-Senecal E, Liu N, Bravin J. Implementing Group CBT for Depression Among Latinos in a Primary Care Clinic. Cogn Behav Pract. 2018 Feb;25(1):135-144. doi: 10.1016/j.cbpra.2017.03.002. PMID 29606848
- [Background] Garcia ME, Ochoa-Frongia L, Moise N, Aguilera A, Fernandez A. Collaborative Care for Depression among Patients with Limited English Proficiency: a Systematic Review. J Gen Intern Med. 2018 Mar;33(3):347-357. doi: 10.1007/s11606-017-4242-4. Epub 2017 Dec 18. PMID 29256085
- [Background] Aguilera A, Ramos Z, Sistiva D, Wang Y, Alegria M. Homework completion via telephone and in-person Cognitive Behavioral Therapy among Latinos. Cognit Ther Res. 2018 Jun;42(3):340-347. Epub 2018 Jan 6. PMID 29725144
- [Background] Aguilera A, Bruehlman-Senecal E, Demasi O, Avila P. Automated Text Messaging as an Adjunct to Cognitive Behavioral Therapy for Depression: A Clinical Trial. J Med Internet Res. 2017 May 8;19(5):e148. doi: 10.2196/jmir.6914. PMID 28483742
- [Background] Avila-Garcia P, Hernandez-Ramos R, Nouri SS, Cemballi A, Sarkar U, Lyles CR, Aguilera A. Engaging users in the design of an mHealth, text message-based intervention to increase physical activity at a safety-net health care system. JAMIA Open. 2019 Oct 11;2(4):489-497. doi: 10.1093/jamiaopen/ooz049. eCollection 2019 Dec. PMID 32025646
- [Background] Nouri SS, Avila-Garcia P, Cemballi AG, Sarkar U, Aguilera A, Lyles CR. Assessing Mobile Phone Digital Literacy and Engagement in User-Centered Design in a Diverse, Safety-Net Population: Mixed Methods Study. JMIR Mhealth Uhealth. 2019 Aug 29;7(8):e14250. doi: 10.2196/14250. PMID 31469083
- [Background] Mohr DC, Lattie EG, Tomasino KN, Kwasny MJ, Kaiser SM, Gray EL, Alam N, Jordan N, Schueller SM. A randomized noninferiority trial evaluating remotely-delivered stepped care for depression using internet cognitive behavioral therapy (CBT) and telephone CBT. Behav Res Ther. 2019 Dec;123:103485. doi: 10.1016/j.brat.2019.103485. Epub 2019 Sep 30. PMID 31634738
- [Background] Mohr DC, Schueller SM, Tomasino KN, Kaiser SM, Alam N, Karr C, Vergara JL, Gray EL, Kwasny MJ, Lattie EG. Comparison of the Effects of Coaching and Receipt of App Recommendations on Depression, Anxiety, and Engagement in the IntelliCare Platform: Factorial Randomized Controlled Trial. J Med Internet Res. 2019 Aug 28;21(8):e13609. doi: 10.2196/13609. PMID 31464192
- [Background] Lattie EG, Ho J, Sargent E, Tomasino KN, Smith JD, Brown CH, Mohr DC. Teens Engaged in Collaborative Health: The Feasibility and Acceptability of an Online Skill-Building Intervention for Adolescents at Risk for Depression. Internet Interv. 2017 Jun;8:15-26. doi: 10.1016/j.invent.2017.02.003. Epub 2017 Mar 2. PMID 28584734
- [Background] Tomasino KN, Lattie EG, Ho J, Palac HL, Kaiser SM, Mohr DC. Harnessing Peer Support in an Online Intervention for Older Adults with Depression. Am J Geriatr Psychiatry. 2017 Oct;25(10):1109-1119. doi: 10.1016/j.jagp.2017.04.015. Epub 2017 May 3. PMID 28571785
- [Background] Mohr DC, Tomasino KN, Lattie EG, Palac HL, Kwasny MJ, Weingardt K, Karr CJ, Kaiser SM, Rossom RC, Bardsley LR, Caccamo L, Stiles-Shields C, Schueller SM. IntelliCare: An Eclectic, Skills-Based App Suite for the Treatment of Depression and Anxiety. J Med Internet Res. 2017 Jan 5;19(1):e10. doi: 10.2196/jmir.6645. PMID 28057609
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Glasgow RE. What does it mean to be pragmatic? Pragmatic methods, measures, and models to facilitate research translation. Health Educ Behav. 2013 Jun;40(3):257-65. doi: 10.1177/1090198113486805. PMID 23709579
- [Background] Castel LD, Williams KA, Bosworth HB, Eisen SV, Hahn EA, Irwin DE, Kelly MA, Morse J, Stover A, DeWalt DA, DeVellis RF. Content validity in the PROMIS social-health domain: a qualitative analysis of focus-group data. Qual Life Res. 2008 Jun;17(5):737-49. doi: 10.1007/s11136-008-9352-3. Epub 2008 May 14. PMID 18478368
- [Background] Hahn EA, Devellis RF, Bode RK, Garcia SF, Castel LD, Eisen SV, Bosworth HB, Heinemann AW, Rothrock N, Cella D; PROMIS Cooperative Group. Measuring social health in the patient-reported outcomes measurement information system (PROMIS): item bank development and testing. Qual Life Res. 2010 Sep;19(7):1035-44. doi: 10.1007/s11136-010-9654-0. Epub 2010 Apr 25. PMID 20419503
- [Background] Enrique A, Mooney O, Salamanca-Sanabria A, Lee CT, Farrell S, Richards D. Assessing the efficacy and acceptability of an internet-delivered intervention for resilience among college students: A pilot randomised control trial protocol. Internet Interv. 2019 Jun 18;17:100254. doi: 10.1016/j.invent.2019.100254. eCollection 2019 Sep. PMID 31304095
- [Background] Chien I, Enrique A, Palacios J, Regan T, Keegan D, Carter D, Tschiatschek S, Nori A, Thieme A, Richards D, Doherty G, Belgrave D. A Machine Learning Approach to Understanding Patterns of Engagement With Internet-Delivered Mental Health Interventions. JAMA Netw Open. 2020 Jul 1;3(7):e2010791. doi: 10.1001/jamanetworkopen.2020.10791. PMID 32678450
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Graham AK, Lattie EG, Mohr DC. Experimental Therapeutics for Digital Mental Health. JAMA Psychiatry. 2019 Dec 1;76(12):1223-1224. doi: 10.1001/jamapsychiatry.2019.2075. No abstract available. PMID 31433448
- [Background] Mohr DC, Cuijpers P, Lehman K. Supportive accountability: a model for providing human support to enhance adherence to eHealth interventions. J Med Internet Res. 2011 Mar 10;13(1):e30. doi: 10.2196/jmir.1602. PMID 21393123
- [Background] Terides MD, Dear BF, Fogliati VJ, Gandy M, Karin E, Jones MP, Titov N. Increased skills usage statistically mediates symptom reduction in self-guided internet-delivered cognitive-behavioural therapy for depression and anxiety: a randomised controlled trial. Cogn Behav Ther. 2018 Jan;47(1):43-61. doi: 10.1080/16506073.2017.1347195. Epub 2017 Jul 20. PMID 28724338
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Ehrhart MG, Aarons GA, Farahnak LR. Assessing the organizational context for EBP implementation: the development and validity testing of the Implementation Climate Scale (ICS). Implement Sci. 2014 Oct 23;9:157. doi: 10.1186/s13012-014-0157-1. PMID 25338781
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- [Background] McMillan D, Gilbody S, Richards D. Defining successful treatment outcome in depression using the PHQ-9: a comparison of methods. J Affect Disord. 2010 Dec;127(1-3):122-9. doi: 10.1016/j.jad.2010.04.030. Epub 2010 May 31. PMID 20569992
- [Background] Manara GC, Ferrari C, Scandroglio R, Rocchi G, Pagani L, De Panfilis G. Characterization of two morphologically distinct Leu-7+ cell subsets with respect to Leu-15 antigen. Evaluation of Leu-15 determinant distribution on both E rosetting and non-adherent non-E rosetting cell populations. Scand J Immunol. 1986 Feb;23(2):225-31. doi: 10.1111/j.1365-3083.1986.tb01961.x. PMID 2419967
- [Background] Paxling B, Lundgren S, Norman A, Almlov J, Carlbring P, Cuijpers P, Andersson G. Therapist behaviours in internet-delivered cognitive behaviour therapy: analyses of e-mail correspondence in the treatment of generalized anxiety disorder. Behav Cogn Psychother. 2013 May;41(3):280-9. doi: 10.1017/S1352465812000240. Epub 2012 May 1. PMID 22717145
- [Background] Carlbring P, Gunnarsdottir M, Hedensjo L, Andersson G, Ekselius L, Furmark T. Treatment of social phobia: randomised trial of internet-delivered cognitive-behavioural therapy with telephone support. Br J Psychiatry. 2007 Feb;190:123-8. doi: 10.1192/bjp.bp.105.020107. PMID 17267928
- [Background] Grol R, Wensing M. What drives change? Barriers to and incentives for achieving evidence-based practice. Med J Aust. 2004 Mar 15;180(S6):S57-60. doi: 10.5694/j.1326-5377.2004.tb05948.x. PMID 15012583
- [Background] DeSantis L, Ugarriza DN. The concept of theme as used in qualitative nursing research. West J Nurs Res. 2000 Apr;22(3):351-72. doi: 10.1177/019394590002200308. PMID 10804897
- [Background] 2016 National Healthcare Quality and Disparities Report. Rockville, MD: Agency for Healthcare Research and Quality; October 2017. AHRQ Pub. No. 17-0001.
- [Background] Escovar, EL. Engagement and premature dropout among Latinx and non-Latinx White patients in a cognitive-behavioral intervention for anxiety. Los Angeles, CA: Psychology, University of California, Los Angeles; 2019. https://escholarship.org/uc/item/3gp4x85h
- [Background] Auntré H, Karen S, Luona L, Peggy C. 2015 APA Survey of Psychology Health Service Providers. American Psychological Association Center for Workforce Studies; 2016
- [Background] Nguyen BP. Identification: Aqualitative study of the experiences of bilingual therapists with their monolinguals and bilingual clients. Psychodynamic Practice: Individuals, Groups and Organisations. 2014;20(4):340-355. DOI: 10.1080/14753634.2014.947168
- [Background] Parks AC, Williams AL, Tugade MM, et al. Testing a scalable web and smartphone based intervention to improve depression, anxiety, and resilience: A randomized controlled trial. International Journal of Wellbeing. 2018;8(2):22-67. DOI:10.5502/ijw.v8i2.745
- [Background] Doherty G, Coyle, D., Sharry J. Engagement with online mental health interventions: an exploratory clinical study of a treatment for depression. Proceedings of the SIGCHI Conference on Human Factors in Computing Systems. 2012; 1421-1430. DOI:10.1145/2207676.2208602
- [Background] Brown CH, Mason WA, Brown EC. Translating the intervention approach into an appropriate research design: The next generation designs for effectiveness and implementation research. In: Sloboda Z, Petras H, eds. Advances in Prevention Science: Defining Prevention Science. New York: Springer; 2014:363-388.
- [Background] Tomasino KN, Noth F, Bardsley LR, Lattie EG, Mohr DC. Intellicare Study Coaching Manual. DigitalHub: Northwestern University;2016.
- [Background] Miranda J, Woo, S., Lagomasino, I., Hepner, K. A., WIseman, S., Munoz, R. F. BRIGHT CBT Depression Group Manuals. http://i4health.paloaltou.edu/manuals/bright-manuals.html. Published 2006. Accessed.
- [Background] Norris AE, Ford K, Bova CA. Psychometrics of a brief acculturation scale for hispanics in a probability sample of urban Hispanic adolescents and young adults. Hispanic J Behav Sci. 1996;18(1):29-38. DOI:10.1177/07399863960181004
- [Background] The MacArthur Foundation's Initiative on Depression and Primary Care. The Macarthur initiative on depression and primary care at Dartmouth and Duke: Depression management toolkit. Hanover, NH: Dartmouth;2004.
- [Background] Berg M, Andersson, G., Rozental, A. Knowledge about treatment, anxiety, and depression in association with internet-based cognitive behavioral therapy for adolescents: Development and initial evaluation of a new test. SAGE Open. 2020;10(1). doi: 10.1177/2158244019899095.
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative research in psychology. 2006;3(2):77-101. DOI: 10.1191/1478088706qp063oa
- [Background] Braun V, Clarke V, Terry G. Thematic analysis. Qual Res Clin Health Psychol. 2014;3(2):77-101.
- [Background] Muhr T. Atlas.ti. In. Berlin: Scientific Software Development; 1997
- [Background] Morse JM, Barrett, M., Mayan, M., Olson, K., & Splers, J. Verification strategies for establishing reliability and validity in qualitative research. International Journal of Qualitative Methods. 2002;1(2):13- 22. DOI: 10.1177/160940690200100202
- [Background] Little RJA, Rubin DB. Statistical Analysis with Missing Data, 2nd Ed. New York: Wiley; 2002
- [Background] Preisser JS, Lohman KK, Craven TE, Wagenknecht LE. Analysis of smoking trends with incomplete longitudinal binary responses. Journal of the American Statistical Association. 2000;95:1021-1031. DOI: 10.1080/01621459.2000.10474299
- [Background] Hill CE, Thompson BJ, Williams EN. A guide to conducting consensual qualitative research. The counseling psychologist. 1997;25(4):517-572. DOI: 10.1177/001100097254001
- [Background] Hill CE, Knox S, Thompson BJ, Williams EN, Hess SA, Ladany N. Consensual qualitative research: An update. Journal of counseling psychology. 2005;52(2):196-205. DOI: 10.1037/0022-0167.52.2.196
- [Background] Auntré H, Karen S, Luona L, Peggy C. 2015 APA Survey of Psychology Health Service Providers. American Psychological Association Center for Workforce Studies; 2016.
- [Background] National Institute for Health and Clinical Excellence (NICE). Computerised cognitive behaviour therapy for depression and anxiety. London: National Institute for Health and Clinical Excellence. 2006. https://www.nice.org.uk/guidance/ta97
- [Derived] Aguilera A, Arevalo Avalos MR, Rosales K, Reyes Y, Hernandez-Ramos R, Ramos G, Garcia E, Hoang T, Ochoa-Frongia L, Fortuna LR, Schueller SM. Effectiveness-implementation hybrid trial of Spanish language, digital cognitive-behavioral therapy (dCBT) intervention for depression and anxiety - protocol for the SUPERA (SUpport from PEeRs to expand Access) study. Contemp Clin Trials. 2024 Feb;137:107422. doi: 10.1016/j.cct.2023.107422. Epub 2023 Dec 24. PMID 38145715

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05746767/Prot_SAP_000.pdf